CLINICAL TRIAL: NCT03134287
Title: Feasibility of Nasogastric Tube Placement on Intubated Patient: Comparison Between Two-Finger Method and Reverse Sellick's Maneuver
Brief Title: Nasogastric Tube Placement on Intubated Patient: Two-Finger Method vs Reverse Sellick's Maneuver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Aida Rosita Tantri SpAn-KA, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes013
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Adult Patient Undergoing Elective Surgery With General Anesthesia and Needs Nasogastric Tube Placement

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- two-finger method (Active Comparator): Those who received nasogastric tube placement by two-finger method
  Interventions: Procedure: two-finger method, reverse sellick's method
- reverse sellick's method (Active Comparator): Those who received nasogastric tube placement by reverse sellick's method
  Interventions: Procedure: two-finger method, reverse sellick's method

INTERVENTIONS:
Procedure: two-finger method, reverse sellick's method — Subjects received nasogastric tube placement by two-finger method; Subjects received nasogastric tube placement by reverse sellick's method

SUMMARY:
The study aimed to compare the efficacy between nasogastric tube placement using Two-Finger Method and Reverse Sellick's Maneuver

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study and randomized into two groups (Two-Finger method group and Reverse Sellick's maneuver group). Intravenous (IV) cannula with isotonic fluid, non-invasive blood pressure monitor, and pulse-oxymetry were set on the subjects in the operation room. Vital signs were recorded. Midazolam 1-2 mg and Fentanyl 2 µg/kg body weight (BW) were given as premedication. Induction was performed using propofol 2-3 µg/kg BW. Rocuronium 0.5mg/kg BW was also given after induction. Two minimum alveolar concentration (MAC) of sevoflurane and 6 liter per minute of oxygen were also given using face mask for 3 minutes until the drugs took effect. Patient were then intubated. Evaluation of airway was performed to exclude the subjects who experienced airway trauma. Estimating the length of nasogastric tube was performed by stretching the nasogastric tube from xyphoid process through nose to the back of the ear. The measured number in cm then added with 15 cm and marked with tape. Nasogastric tube and the selected nostril then covered in gel sufficiently. The Two-Finger method group was placed with nasogastric tube using two-finger method, before the procedure, the endotracheal tube cuff was deflated first. And then the nasogastric tube was inserted into the selected nostril perpendicularly using dominant hand. The non-dominant hand (index and middle finger) was inserted to the base of oropharynx until the nasogastric tube was felt , and the the nasogastric tube was fixated in the middle position and the base of pharynx, as nearest as possible from esophagus, while the dominant hand pushed the nasogastric tube until it reached the mark. The reverse Sellick's maneuver group's endotracheal tube was also deflated before the procedure. The nasogastric tube was inserted into the selected nostril perpendicularly using dominant hand and pushed gently until it reached the first resistance in nasopharynx. Reverse Sellick's maneuver was performed using non-dominant hand, done by grabbing thyroid cartilage upward and elevated the larynx anteriorly, while the dominant hand kept pushing the nasogastric tube gently until it reached the mark. Evaluation whether or not the nasogastric tube was properly placed was using the auscultation method in the epigastric region and inserting air through catheter tip. Time and complications occurred during procedure were recorded. And the nasogastric tube was fixated if it was successfully inserted.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-60 years old, with American Society of Anesthesiologists (ASA) physical status of I-III who were planned to undergo any elective surgery at operating room in general anesthesia and needed nasogastric tube placement
* subjects had been explained about the study, and agreed to enroll and have signed the informed consent form

Exclusion Criteria:

* Subjects with possibility of difficult airway
* multiple fracture in the head
* craniofacial, airway, esophagus, and neck abnormality

Drop out Criteria:

* Subjects who experience airway trauma during intubation or allergic reaction due to drugs used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Successful rate | Day 1
  Successful rate on nasogastric tube placement in first attempt

SECONDARY OUTCOMES:
Time | Day 1
  Time needed to insert the nasogastric tube
Complications | Day 1
  Complications occurred during procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sinha PK, Koshy T. Reverse Sellick's maneuver for transesophageal echocardiographic probe placement. J Cardiothorac Vasc Anesth. 2007 Aug;21(4):626-8. doi: 10.1053/j.jvca.2006.10.010. Epub 2007 Jan 9. No abstract available. PMID 17678806
- [Background] Ratzlaff HC, Heaslip JE, Rothwell ES. Factors affecting nasogastric tube insertion. Crit Care Med. 1984 Jan;12(1):52-3. doi: 10.1097/00003246-198401000-00014. PMID 6690206
- [Background] Ozer S, Benumof JL. Oro- and nasogastric tube passage in intubated patients: fiberoptic description of where they go at the laryngeal level and how to make them enter the esophagus. Anesthesiology. 1999 Jul;91(1):137-43. doi: 10.1097/00000542-199907000-00022. PMID 10422939
- [Background] Kirtania J, Ghose T, Garai D, Ray S. Esophageal guidewire-assisted nasogastric tube insertion in anesthetized and intubated patients: a prospective randomized controlled study. Anesth Analg. 2012 Feb;114(2):343-8. doi: 10.1213/ANE.0b013e31823be0a4. Epub 2011 Nov 21. PMID 22104075
- [Background] Agarwal A, Gaur A, Sahu D, Singh PK, Pandey CK. Nasogastric tube knotting over the epiglottis: a cause of respiratory distress. Anesth Analg. 2002 Jun;94(6):1659-60, table of contents. doi: 10.1097/00000539-200206000-00056. PMID 12032048
- [Background] Cataldi-Betcher EL, Seltzer MH, Slocum BA, Jones KW. Complications occurring during enteral nutrition support: a prospective study. JPEN J Parenter Enteral Nutr. 1983 Nov-Dec;7(6):546-52. doi: 10.1177/0148607183007006546. PMID 6418910
- [Background] Noguchi T, Shiga Y, Koga K, Shigematsu A. A method to improve a gas leak on mask ventilation in the patient with a nasogastric tube. Anesthesiology. 2001 Mar;94(3):545. doi: 10.1097/00000542-200103000-00041. No abstract available. PMID 11374627
- [Background] Appukutty J, Shroff PP. Nasogastric tube insertion using different techniques in anesthetized patients: a prospective, randomized study. Anesth Analg. 2009 Sep;109(3):832-5. doi: 10.1213/ane.0b013e3181af5e1f. PMID 19690254
- [Background] Mahajan R, Gupta R, Sharma A. Role of neck flexion in facilitating nasogastric tube insertion. Anesthesiology. 2005 Aug;103(2):446-7. doi: 10.1097/00000542-200508000-00034. No abstract available. PMID 16052133
- [Background] Chun DH, Kim NY, Shin YS, Kim SH. A randomized, clinical trial of frozen versus standard nasogastric tube placement. World J Surg. 2009 Sep;33(9):1789-92. doi: 10.1007/s00268-009-0144-x. PMID 19626360
- [Background] Moharari RS, Fallah AH, Khajavi MR, Khashayar P, Lakeh MM, Najafi A. The GlideScope facilitates nasogastric tube insertion: a randomized clinical trial. Anesth Analg. 2010 Jan 1;110(1):115-8. doi: 10.1213/ANE.0b013e3181be0e43. Epub 2009 Oct 27. PMID 19861362
- [Background] Perel A, Ya'ari Y, Pizov R. Forward displacement of the larynx for nasogastric tube insertion in intubated patients. Crit Care Med. 1985 Mar;13(3):204-5. doi: 10.1097/00003246-198503000-00013. PMID 3971730
- Available data/document: Textbook — http://onlinelibrary.wiley.com/doi/10.1111/j.1742-6723.2004.00655.x/full — Samuels LE, Roberts JR, Hedges JR. Nasogastric and Feeding Tube Placement, In: Clinical Procedures in Emergency Medicine. 4th ed. WB Saunders; 2004. p784-804.
- Available data/document: Textbook — https://books.google.co.id/books?id=ooH1nH81_h4C&pg=PR4&lpg=PR4&dq=Irwin+and+Rippe%27s+Intensive+Care+Medicine+2008&source=bl&ots=43X9QRBshe&sig=Y3ycuRyss2vYHzN3q0WFtrSdPRM&hl=en&sa=X&ved=0ahUKEwjk_6TIo8LTAhWMvY8KHSvTDo8Q6AEIRzAG#v=onepage&q=Irwin%20and%20Rippe's%20Intensive%20Care%20Medicine%202008&f=false — Irwin RS, Rippe JM. Irwin and Rippe's Intensive Care Medicine: Endoscopic Placement of Feeding Tubes. 6th ed. Lippincott Williams & Wilkins; 2008. p145-150.
- Available data/document: Textbook — https://books.google.co.id/books/about/The_ICU_Book.html?id=OWEmVx9MS74C&redir_esc=y — Marino PL. Enteral Tube Feeding. In: The ICU Book. 3rd ed. Lippincott Williams & Wilkins; 2007. p842-855.